CLINICAL TRIAL: NCT05889897
Title: Prevalence, Risk Factors and Outcomes of Vascular Thromboembolism in Children Attending Assuit University Hospital
Brief Title: Prevalence, Risk Factors and Outcomes of Pediatric Vascular Thrombosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Doaa Sayed Shaker Ahmed, principle investigator, Assiut University
Other Study IDs: pediatric vascular thrombosis
Record Dates: First submitted 2023-03-26; First posted 2023-06-05 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Vascular Thrombosis
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

SUMMARY:
This study is aimed to identify the prevalence, risk factors and outcomes of children with either venous or arterial thromboembolism admitted to children hospital Assiut University aiming at early detection and avoidance of catastrophic complications .

DETAILED DESCRIPTION:
Thrombosis is a blood clot that develops within veins or sometimes arteries in the body.

Occur most commonly in the inferior and superior vena cava, their major tributaries, the deep veins of the extremities, the splanchnic veins, as well as the cerebral venous sinuses.

The incidence of venous thromboembolism (VTE) increases with age. In the pediatric population (0-18 years) the incidence is approximately 0.7-2.1 cases per 100,000 children,1-3 while in the adult population the incidence is 100-150 per 100,000.4

Risk factors include the presence of central venous lines, trauma, major surgery followed by bedrest, immobilization, infection (cellulitis, osteomyelitis, phlebitis), cancer chemotherapy, inflammatory bowel disease, nephrotic syndrome, obesity, dehydration, and total parenteral nutrition.

Patients with vascular thromboembolism present with various symptoms depending on site of thrombosis , symptoms include swelling, redness, pain , low-grade fever In cases that develop pulmonary embolism they experience chest pain and shortness of breath that begin suddenly

Diagnosis of vascular thromboembolism include combination of signs and symptoms together with laboratory investigations that include routine lab investigations, D-dimer , protein s , protein C and antithrombin lll also imaging studies as Doppler US , MSCT with angiography and MRV

Vascular thrombosis mainly treated with anticoagulant therapy with subcutaneous injection of low molecular weight heparin These medications prevent the clot from growing and decrease the risk of its breaking apart and causing further complications Other treatments may include wearing compression stockings and applying warm packs to improve blood flow and pain caused by the clot

ELIGIBILITY:
Inclusion Criteria :

* Age : From 1day to 18 years.
* Sex : Both genders.
* Confirmed diagnosed cases, either Symptomatic or asymptomatic venous and arterial thromboembolism established by an imaging study.
* All patients admitted to the different units of children hospital including surgical unit.

Exclusion Criteria :

* Age more than 18 years.
* Patient Known to have Sickle cell disease.

Ages: 1 Day to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: 15 infant aged from 1 day to 18 years with vascular thrombosis
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Number of pediatrics with vascular thrombosis | baseline
  This study is aimed to identify the prevalence of children with either venous or arterial thromboembolism admitted to children hospital Assiut University aiming at early detection and avoidance of catastrophic complications
Number of risk factors of pediatric vascular thrombosis | Baseline
  This study is aimed to identify risk factors of children with either venous or arterial thromboembolism admitted to children hospital Assiut University aiming at early detection and avoidance of catastrophic complications

CONTACTS AND LOCATIONS:
Overall Officials: Maher Mokhtar, Prof, Principal Investigator — Assiut University; Mervat Amin, Assist Prof, Principal Investigator — Assiut University